CLINICAL TRIAL: NCT03596866
Title: A Phase 3 Randomized Open-label Study of Brigatinib (ALUNBRIG®) Versus Alectinib (ALECENSA®) in Advanced Anaplastic Lymphoma Kinase-Positive Non-Small-Cell Lung Cancer Patients Who Have Progressed on Crizotinib (XALKORI®)
Brief Title: A Study of Brigatinib Compared to Alectinib in Adults With Non-Small-Cell Lung Cancer
Acronym: ALTA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brigatinib-3001; 2018-001957-29 (EudraCT Number)
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: ALK+ Advanced NSCLC
Keywords: Drug Therapy
MeSH Terms: interventions — brigatinib; alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brigatinib (Experimental): Participants were administered brigatinib 90 milligrams (mg), tablets, orally, once daily (QD) for 7 days, followed by brigatinib 180 mg, tablets, orally, QD until objective disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as assessed by the investigator, or intolerable toxicity, or up to 63.47 months.
  Interventions: Drug: Brigatinib
- Alectinib (Active Comparator): Participants were administered alectinib 600 mg, capsules, orally, twice daily (BID) until objective disease progression per RECIST v1.1, as assessed by the investigator, or intolerable toxicity, or up to 59.83 months.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib Tablets.
  Other Names: Alunbrig
  Arms: Brigatinib
Drug: Alectinib — Alectinib Capsules.
  Other Names: Alecensa
  Arms: Alectinib

SUMMARY:
Brigatinib is a medicine that binds to the surface of tumor cells in some cancers and delivers a dose of chemotherapy directly to the tumor. In this study, participants will be people with non-small-cell lung cancer (NSCLC for short). The main aim of the study is to learn if brigatinib stops the tumors from growing, or if the tumors have shrunk or disappeared, compared to a medicine called alectinib.

At the first visit, the study doctor will check who can take part. Participants who can take part will be picked for 1 of 2 treatments by chance:

* Brigatinib tablets
* Alectinib capsules

All participants will take brigatinib or alectinib at about the same time every day. They will continue with treatment throughout the study unless their cancer gets worse, they have side effects from the treatment, they leave the study for certain reasons, or the study is stopped.

After stopping treatment, participants will visit the study clinic for a check-up 30 days later.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib. Brigatinib has been demonstrated to benefit people with anaplastic lymphoma kinase-positive (ALK+) NSCLC.

The comparator drug is called alectinib. Alectinib has been demonstrated to benefit people with ALK+ NSCLC. Both drugs belong to a class of drugs called anaplastic lymphoma kinase (ALK) inhibitors. Both drugs are taken by mouth. Both drugs are approved by the United States Food and Drug Administration (US FDA).

The study will enroll approximately 246 participants. Participants will be randomly assigned (by chance, like flipping a coin) in 1:1 ratio to one of the two treatment groups:

* Brigatinib
* Alectinib

All participants will be asked to take brigatinib or alectinib at the same time each day throughout the study. For each participant eligible to continue in the study and to facilitate the remaining participants from Brigatinib-2002 (NCT03535740) to have continued treatment access, the study extension phase may be initiated for participants to continue receiving their randomized study treatment (i.e., brigatinib or alectinib) until they meet at least one of the treatment discontinuation criteria.

This multi-center trial will be conducted in the United States, Argentina, Austria, Canada, Chile, China, Croatia, France, Germany, Greece, Hong Kong, Italy, Mexico, Romania, Russia, South Korea, Spain, Sweden, Taiwan, and Thailand. The overall time to participate in this study is 5 years. Participants will make multiple visits to the clinic, and 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
2. Have histologically or cytologically confirmed stage IIIB (locally advanced or recurrent) or stage IV NSCLC.
3. Must meet one of the following criteria:

   * Have documentation of ALK rearrangement by a positive result from the Vysis ALK Break-Apart fluorescence in situ hybridization (FISH) Probe Kit or the Ventana ALK (D5F3) CDx Assay or Foundation Medicine's FoundationOne CDx.
   * Have documented ALK rearrangement by a different test and be able to provide tumor sample to the central laboratory. (Note: central laboratory ALK rearrangement testing results are not required to be obtained before randomization).
4. Had PD while on crizotinib, as assessed by the investigator or treating physician except for participants previously participating in the Brigatinib-2002 study (Note: crizotinib does not need to be the last therapy a participant received. The participant may have received chemotherapy as his/her last therapy).
5. Treatment with crizotinib for at least 4 weeks before progression except for participants previously participating in the Brigatinib-2002 study.
6. Have had no other ALK inhibitor other than crizotinib except for participants previously participating in the Brigatinib-2002 study.
7. Have had no more than 2 prior regimens of systemic anticancer therapy (other than crizotinib) in the locally advanced or metastatic setting. Note: a systemic anticancer therapy regimen will be counted if it is administered for at least 1 complete cycle. A new anticancer agent used as maintenance therapy will be counted as a new regimen. Neoadjuvant or adjuvant systemic anticancer therapy will be counted as a prior regimen if disease progression/recurrence occurred within 12 months upon completion of this neoadjuvant or adjuvant therapy. (Systemic therapy followed by maintenance therapy will be considered as one regimen if the maintenance therapy consists of a drug or drugs that were used in the regimen that immediately preceded maintenance).
8. Have at least 1 measurable (that is, target) lesion per RECIST v1.1.
9. Have recovered from toxicities related to prior anticancer therapy to national cancer institute common terminology criteria for adverse events (NCI CTCAE) version 4.03 grade less than or equal to (<=)1. (Note: treatment-related alopecia or peripheral neuropathy that are grade greater than (>) 1 are allowed, if deemed irreversible).
10. Have adequate organ function, at the time of initial screening, except for participants previously participating in the Brigatinib-2002 study as determined by:

    * Total bilirubin <=1.5 times the upper limit of normal (ULN).
    * Estimated glomerular filtration rate greater than equal to (>=) 30 milliliter per minute (mL/min)/1.73 square meter [m^2], using the modification of diet in renal disease equation.
    * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) <=2.5*ULN; <=5*ULN is acceptable if liver metastases are present.
    * Serum lipase <=1.5*ULN.
    * Platelet count >=75*10^9 per liter [/L].
    * Hemoglobin >=9 gram per deciliter (g/dL).
    * Absolute neutrophil count >=1.5*10^9 / L.
11. Suitable venous access for study-required blood sampling (that is, including pharmacokinetic [PK] and laboratory safety tests).

Exclusion Criteria:

1. Had participated in the control (crizotinib) arm of Study AP26113-13-301 (ALTA 1L) [NCT02737501].
2. Had received crizotinib within 7 days before randomization.
3. Have a history or presence at baseline of pulmonary interstitial disease, drug related pneumonitis, or radiation pneumonitis.
4. Have uncontrolled hypertension. Participants with hypertension should be under treatment for control of blood pressure upon study entry.
5. Had received systemic treatment with strong cytochrome P-450 (CYP) 3A inhibitors, moderate CYP3A inhibitors, strong CYP3A inducers, or moderate CYP3A inducers within 14 days before randomization.
6. Treatment with any investigational systemic anticancer agents within 14 days or 5 half-lives, whichever is longer, before randomization.
7. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated nonmelanoma skin cancer or cervical cancer in situ; definitively treated nonmetastatic prostate cancer; or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
8. Had received chemotherapy or radiation therapy within 14 days before randomization except for stereotactic radiosurgery (SRS) or stereotactic body radiation therapy.
9. Had received antineoplastic monoclonal antibodies within 30 days of randomization.
10. Had major surgery within 30 days of randomization. Minor surgical procedures, such as catheter placement or minimally invasive biopsies, are allowed.
11. Have symptomatic CNS metastases (parenchymal or leptomeningeal) at screening (participants with asymptomatic brain metastases or participants who have stable symptoms and did not require an increased dose of corticosteroids to control symptoms within 7 days before randomization will be enrolled). Note: If a participant has worsening neurological symptoms or signs due to CNS metastasis, the participant needs to complete local therapy and be neurologically stable (with no requirement for an increasing dose of corticosteroids or use of anticonvulsants) for 7 days before randomization.
12. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Participants with leptomeningeal disease and without cord compression are allowed.
13. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to the following:

    * Myocardial infarction within 6 months before randomization.
    * Unstable angina within 6 months before randomization.
    * New York Heart Association Class III or IV heart failure within 6 months before randomization.
    * History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician.
    * Any history of clinically significant ventricular arrhythmia.
14. Had cerebrovascular accident or transient ischemic attack within 6 months before first dose of study drug.
15. Have malabsorption syndrome or other gastrointestinal illness or condition that could affect oral absorption of the study drug.
16. Have an ongoing or active infection, including but not limited to, the requirement for intravenous antibiotics.
17. Have a known history of human immunodeficiency virus (HIV) infection. Testing is not required in the absence of history.
18. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection. Testing is not required in the absence of history.
19. Any serious medical condition or psychiatric illness that could, in the investigator's opinion, potentially compromise participant safety or interfere with the completion of treatment according to this protocol.
20. Have a known or suspected hypersensitivity to brigatinib or alectinib or their excipients.
21. Life-threatening illness unrelated to cancer.
22. Female participants who are lactating and breastfeeding.
23. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (113):
- United States (4):
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University Cancer and Blood Center, Athens, Georgia
  - New York Oncology Hematology - Albany Medical Center, Albany, New York
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (3):
  - Centro Para la Atencion Integral del Paciente Oncologico, San Miguel de Tucumán, Tucumán Province
  - Sanatorio Duarte Quiros, Córdoba
  - Centro Oncologico Riojano Integral, La Rioja
- Klinikum Klagenfurt Am Worthersee, Klagenfurt, Carinthia, Austria
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Toronto University Health Network, Toronto, Ontario
- Centro de Investigacion Clinica Bradford Hill, Recoleta, Santiago Metropolitan, Chile
- China (14):
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital - East, Beijing, Beijing Municipality
  - Peking University Cancer Hospital/Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The 307th Hospital of Chinese Peoples Liberation Army, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Harbin Medical University - The 3rd Affiliated Hospital of HMU, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jilin Provincial Cancer Hospital (Changchun Cancer Hospital), Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Chang Gung Memorial Hospital Linkou Branch, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
- Croatia (5):
  - Fudan University Shanghai Cancer Center, Dubrovnik, Dubrovnik-Neretva County
  - Opca bolnica Dubrovnik, Dubrovnik, Dubrovnik-Neretva County
  - General Hospital Pula, Pula
  - Klinicki bolnicki centar Sestre milosrdnice, Zagreb
  - Klinika za Pulmologiju, Zagreb
- France (9):
  - Hopital Haut-Leveque, Pessac, Aquitaine
  - Hopital Albert Michallon, Grenoble, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Toulouse- Hopital Larrey, Toulouse, Midi-pyrenees
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Intercommunal Toulon - La Seyne Sur Mer, Toulon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Intercommunal de Creteil, Créteil, Île-de-France Region
  - Fudan University Shanghai Cancer Center, Créteil, Île-de-France Region
  - Hopital Foch, Suresnes, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (3):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Asklepios Fachkliniken Munchen-Gauting, Gauting, Bavaria
  - Klinikum Kempten-Oberallgau, Immenstadt im Allgäu, Bavaria
- Greece (6):
  - University General Hospital of Athens Attikon, Athens, Attica
  - Iaso General Hospital, Cholargós, Attica
  - General Oncology Hospital of Kifisia Oi Agioi Anargiroi, Nea Kifissia, Attica
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki, Macedonia
  - University General Hospital of Larissa, Larissa, Thessaly
  - Sotiria General Hospital for Respiratory Diseases of Attica, Athens
- Hong Kong (5):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan, Eastern District
  - Humanity and Health Research Centre, Central
  - Queen Mary Hospital, Hong Kong
  - Hong Kong United Oncology Centre, Kowloon
  - Princess Margaret Hospital, Kowloon
- Italy (7):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-cesena
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Ospedale Santa Maria delle Croci, Ravenna
- Mexico (2):
  - Medica Sur, Mexico City, Mexico City
  - Centro de Investigacion Medica Aguascalientes, Aguascalientes
- Romania (4):
  - Institutul Oncologic Prof. Dr. Ion Chiricu, Cluj-Napoca, Cluj
  - Oncocenter- Oncologie Clinica, Timișoara, Timiș County
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu Bucaresti, Bucharest
  - Centrul de oncologie Euroclinic, Iași
- Russia (13):
  - State Institution of Healthcare Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arkhangelr
  - Euromedservice, Saint Petersburg, Sankt-Peterburg
  - Saint Petersburg Clinical Scientific and Practical Center of Specialized Types of Medical Aid, Saint Petersburg, Sankt-Peterburg
  - Clinica Ultra Sound Diagnostic 4D, Pyatigorsk, Stavropol Kray
  - Irkutsk Regional Oncology Center, Irkutsk
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - VitaMed, Moscow
  - State Budget Institution National Medical Research Center of Radiology of the Ministry of Heal, Moscow
  - Moscow City Oncology Hospital Number 62, Moscow
  - Omsk Regional Clinical Oncologic Dispensary, Omsk
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Center of Palliative Medicine - Devita, Saint Petersburg
  - Saint Petersburg State Healthcare Institution Municipal Clinical Oncology Dispensary, Saint Petersburg
- South Korea (10):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Ulsan University Hospital, Ulsan, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Teresa Herrera - Materno Infantil, A Coruña, LA Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (2):
  - Karolinska Universitetssjukhuset - Solna, Solna, Stockholm County
  - Uppsala Akademiska Sjukhus, Uppsala
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok, Bangkok Metropolis
  - Phramongkutklao Hospital, Bangkok, Bangkok Metropolis
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Yang JC, Liu G, Lu S, He J, Burotto M, Ahn MJ, Kim DW, Liu X, Zhao Y, Vincent S, Yin J, Ma X, Lin HM, Popat S. Brigatinib Versus Alectinib in ALK-Positive NSCLC After Disease Progression on Crizotinib: Results of Phase 3 ALTA-3 Trial. J Thorac Oncol. 2023 Dec;18(12):1743-1755. doi: 10.1016/j.jtho.2023.08.010. Epub 2023 Aug 12. PMID 37574132
- [Derived] Popat S, Liu G, Lu S, Song G, Ma X, Yang JC. Brigatinib vs alectinib in crizotinib-resistant advanced anaplastic lymphoma kinase-positive non-small-cell lung cancer (ALTA-3). Future Oncol. 2021 Nov;17(32):4237-4247. doi: 10.2217/fon-2021-0608. Epub 2021 Aug 23. PMID 34423676
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b601c4db2bf003ab493af

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 19 April 2019 to 18 September 2024.
Pre-assignment Details: Participants with anaplastic lymphoma kinase positive (ALK+) non-small-cell lung cancer (NSCLC) who had progressed on crizotinib were administered either brigatinib or alectinib in this study.
Period: Overall Study
Arm/Group | Brigatinib | Alectinib
Started | 125 | 123
Completed | 3 | 6
Not Completed | 122 | 117
Not completed — Site terminated by Sponsor | 64 | 65
Not completed — Death | 37 | 24
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Missing | 0 | 6
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Reason Not Specified | 14 | 13

BASELINE CHARACTERISTICS:
Population: Full Analysis Set(FAS) included all participants randomized to each regimen regardless of whether they were ALK+ by an Food and Drug Administration(FDA) approved test (Vysis ALK Break Apart fluorescence in situ hybridization(FISH) Probe Kit, Ventana ALK (D5F3) Companion Diagnostics (CDx) Assay, Foundation Medicine's FoundationOne CDx) or a local test other than FISH and immunohistochemistry, or whether they received study drug or adhered to the assigned dose.
Groups:
- Brigatinib: Participants were administered brigatinib 90 mg, tablets, orally, QD for 7 days, followed by brigatinib 180 mg, tablets, orally, QD until objective disease progression per RECIST v1.1, as assessed by the investigator, or intolerable toxicity, or up to 33.8 months.
- Alectinib: Participants were administered alectinib 600 mg, capsules, orally, BID until objective disease progression per RECIST version 1.1, as assessed by the investigator, or intolerable toxicity, or up to 33.8 months.
- Total: Total of all reporting groups
Arm/Group | Brigatinib | Alectinib | Total
Number analyzed (Participants) | 125 | 123 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (12.17) | 52.9 (13.53) | 53 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 68 | 135
  Male | 58 | 55 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 21
  Not Hispanic or Latino | 116 | 106 | 222
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 74 | 66 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 50 | 52 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Blinded Independent Review Committee (BIRC) Per RECIST v1.1
Description: PFS is defined as the time interval from the date of randomization until the first date at which disease progression is objectively documented via RECIST v1.1 by BIRC, or death due to any cause, whichever occurs first, in the full analysis set. PFS was censored for participants without documented disease progression or death at the last valid tumor response assessment.
Time Frame: Up to 33.8 months
Population: FAS included all participants randomized to each regimen regardless of whether they were ALK+ by an FDA approved test (Vysis ALK Break Apart FISH Probe Kit, Ventana ALK (D5F3) CDx Assay, Foundation Medicine's FoundationOne CDx) or a local test other than FISH and immunohistochemistry, or whether they received study drug or adhered to the assigned dose.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Brigatinib: Participants were administered brigatinib 90 mg, tablets, orally, QD for 7 days, followed by brigatinib 180 mg, tablets, orally, QD until objective disease progression per RECIST v1.1, as assessed by the investigator, or intolerable toxicity, or up to 63.47 months.
- Alectinib: Participants were administered alectinib 600 mg, capsules, orally, BID until objective disease progression per RECIST v1.1, as assessed by the investigator, or intolerable toxicity, or up to 59.83 months.
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 125 | 123
months | 19.253 [15.671 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to censoring. | 19.187 [12.879 to NA] — The upper limit of 95% CI was not estimable due to censoring.
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; Test type: Superiority; p = 0.8672, 2-sided Stratified Log-rank Test — P-value from a 2-sided stratified log-rank test using the stratification factors: presence of intracranial central nervous system (CNS) metastases at baseline, and best prior response to crizotinib therapy as assessed by the investigator; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.658 to 1.424] — The hazard ratio was obtained using the stratified Cox regression model with the same stratification factors

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from the date of randomization until death due to any cause in the full analysis set. OS was censored on the date of last contact for those participants who are alive.
Time Frame: Up to 64 months
Population: FAS included all participants randomized to each regimen regardless of whether they are ALK+ by an FDA approved test (Vysis ALK Break Apart FISH Probe Kit, Ventana ALK (D5F3) CDx Assay, Foundation Medicine's FoundationOne CDx) or a local test other than FISH and immunohistochemistry, or whether they receive study drug or adhere to the assigned dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 125 | 123
months | NA [38.472 to NA] — The median and upper limit of 95% CI was not estimable due to low number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; Test type: Superiority; p = 0.0713, Log Rank — P-value was based on a 2-sided stratified log-rank test using the stratification factors: presence of intracranial CNS metastases at baseline and best prior response to crizotinib therapy as assessed by the investigator; Hazard Ratio (HR) = 1.592, 95% CI 2-sided [0.956 to 2.652] — The HR was obtained using the stratified Cox regression model with the same stratification factors

3. Secondary Outcome: PFS as Assessed by Investigator Per RECIST v1.1
Description: PFS is defined as the time interval from the date of randomization until the first date at which disease progression is objectively documented via RECIST v1.1 by investigator, or death due to any cause, whichever occurs first, in the full analysis set. PFS was censored for participants without documented disease progression or death at the last valid tumor response assessment.
Time Frame: Up to 33.8 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 125 | 123
months | 16.789 [10.940 to 19.417] | 16.591 [13.602 to 27.565]
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; Test type: Superiority; p = 0.2501, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.232, 95% CI 2-sided [0.862 to 1.761] — The HR was obtained using the stratified Cox regression model with the same stratification factors

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BIRC and Investigator Per RECIST v1.1
Description: ORR is defined as the percentage of the participants who are confirmed to have achieved complete response (CR) or partial response (PR), using RECIST v1.1 after the initiation of study treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 33.8 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 125 | 123
percentage of participants
  BIRC Assessed | 52.0 [42.9 to 61.0] | 61.0 [51.8 to 69.6]
  Investigator Assessed | 40.8 [32.1 to 49.9] | 56.1 [46.9 to 65.0]
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; BIRC Assessed; Test type: Superiority; p = 0.1555, Cochran-Mantel-Haenszel — P-value was from a Cochran-Mantel-Haenszel test stratified by the stratification factors: presence of intracranial CNS metastases at baseline and best prior response to crizotinib therapy as assessed by the investigator; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.42 to 1.15] — Odds ratio stratified by the stratification factors: presence of intracranial CNS metastases at baseline and best prior response to crizotinib therapy as assessed by the investigator
Statistical Analysis 2: Comparison: Brigatinib vs Alectinib; Investigator Assessed; Test type: Superiority; p = 0.0169, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.33 to 0.90] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Duration of Response (DOR) as Assessed by BIRC and Investigator Per RECIST v1.1
Description: DOR is defined as the time interval from the time that the measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that the progressive disease (PD) is objectively documented or death, as assessed by the investigator and BIRC, using RECIST v1.1. Participants who did not progress or died, were censored at the last tumor assessment date prior to receiving subsequent anticancer therapy.
Time Frame: Up to 33.8 months
Population: FAS=all participants randomized to each regimen regardless of whether they are ALK+ by an FDA approved test (Vysis ALK Break Apart FISH Probe Kit, Ventana ALK (D5F3) CDx Assay, Foundation Medicine's FoundationOne CDx) or a local test other than FISH and immunohistochemistry, or whether they receive study drug or adhere to the assigned dose. N=number of participants with data available for analysis. n=number of participants with data available for analysis at specified categories.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 78 | 88
months
  BIRC Assessed: number analyzed (Participants) | 65 | 75
  BIRC Assessed | 17.544 [14.784 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events. | 20.205 [12.649 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events.
  Investigator Assessed: number analyzed (Participants) | 51 | 69
  Investigator Assessed | 17.511 [11.335 to 23.031] | 19.614 [14.226 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events.

6. Secondary Outcome: Time to Response as Assessed by Investigator and BIRC Per RECIST v1.1
Description: Time to response is defined as the time interval from randomization until the initial observation of CR or PR, as assessed by the investigator and BIRC, using RECIST v1.1. Time to response will be summarized using descriptive statistics in participants with confirmed objective response.
Time Frame: Up to 33.8 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 78 | 88
months
  BIRC Assessed: number analyzed (Participants) | 65 | 75
  BIRC Assessed | 1.873 [1.64 to 16.49] | 1.840 [1.41 to 16.56]
  Investigator Assessed: number analyzed (Participants) | 51 | 69
  Investigator Assessed | 1.873 [1.61 to 14.00] | 1.873 [1.41 to 10.87]

7. Secondary Outcome: Confirmed Intracranial Objective Response Rate (iORR) as Assessed by BIRC Per Modified RECIST v1.1
Description: Confirmed iORR, as assessed by the BIRC, is defined as the percentage of the participants who have achieved CR or PR in the central nervous system (CNS) per a modification RECIST v1.1 after the initiation of study treatment in participants with CNS metastases at baseline. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 33.8 months
Population: Measurable iCNS disease population included all participants in the full analysis population determined by the BIRC to have had at least 1 measurable iCNS tumor lesion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 30 | 31
percentage of participants | 73.3 [54.1 to 87.7] | 67.7 [48.6 to 83.3]
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; Test type: Superiority; p = 0.6246, Cochran-Mantel-Haenszel — P-value was from a Cochran-Mantel-Haenszel test stratified by best prior response to crizotinib therapy as assessed by the investigator at randomization per IXRS; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.44 to 3.84] — Odds ratio was stratified by best prior response to crizotinib therapy as assessed by the investigator at randomization per IXRS

8. Secondary Outcome: Intracranial Duration of Response (iDOR) as Assessed by the BIRC Per Modified RECIST v1.1
Description: iDOR, as assessed by the BIRC per modified RECIST v1.1, is defined as the time interval from the time that the measurement criteria are first met for CR or PR in the CNS (whichever is first recorded) until the first date that the PD in the CNS is objectively documented or death. Participants who did not progress or died, were censored at the last iCNS tumor assessment date prior to receiving subsequent anticancer therapy.
Time Frame: Up to 33.8 months
Population: Measurable iCNS disease population included all participants in the full analysis population determined by the BIRC to have had at least 1 measurable iCNS tumor lesion. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 22 | 21
months | 17.413 [7.425 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events. | NA [5.552 to NA] — The median and upper limit of 95% CI were not estimable due to low number of participants with events.

9. Secondary Outcome: Cumulative Incidence of Intracranial Disease Progression (iPD) as Assessed by BIRC Per Modified RECIST v1.1
Description: Time to iPD as assessed by the BIRC,is defined as time interval from date of randomization until first date at which iPD is objectively documented via a modification of RECIST v1.1 without prior systemic progression (PD) or death. Time to iPD was analyzed within a competing risk framework (with systemic progression and death as the competing risks) by estimating the cumulative incidence function (CIF) within each arm. The CIF is a function of time, and indicates the probability of an event (e.g. iPD without prior PD or death) occurring by the specified time. The estimated CIFs were analyzed using Grey's Test and the estimated probability of CIFs is reported at pre-specified landmark times (6, 12, 18 and 24 months).
Time Frame: 6, 12, 18 and 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 125 | 123
probability
  6 months | 0.115 [0.064 to 0.182] | 0.076 [0.037 to 0.133]
  12 months | 0.218 [0.144 to 0.302] | 0.171 [0.107 to 0.247]
  18 months | 0.305 [0.211 to 0.404] | 0.209 [0.135 to 0.293]
  24 months | 0.388 [0.274 to 0.500] | 0.248 [0.161 to 0.344]
Statistical Analysis 1: Comparison: Brigatinib vs Alectinib; Test type: Superiority; p = 0.0778, Gray's Test — P-value from a 2-sided stratified Gray's test using the stratification factors (at randomization per IxRS): presence of intracranial CNS metastases at baseline, and best prior response to crizotinib therapy as assessed by the investigator; P-value is for the event type: Intracranial Disease Progression without Prior Systemic Progression or Death

10. Secondary Outcome: Health-Related Quality of Life (HRQOL) From European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 v3.0) Score
Description: EORTC QLQ-C30 incorporates 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status scale, higher scores represent better quality of life (QOL); for the symptom scales, lower scores represent better QOL.
Time Frame: Up to 33.8 months
Population: The patient-reported outcome (PRO) analysis set included all participants with baseline and at least 1 post-baseline PRO measurement in the full analysis set. Overall number analyzed is the number of participants with data available for analysis of this outcome measure at end of treatment visit.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 37 | 41
score on a scale | 86.15 [35.9 to 100.0] | 84.74 [36.6 to 100.0]

11. Secondary Outcome: HRQOL From EORTC QLQ- Lung Cancer (LC) 13
Description: HRQOL scores were assessed with European Organization for Research and Treatment (EORTC), its lung cancer module QLQ-LC13. QLQ-LC13 contains 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Subscales were scored on a range of 0 to 100. Higher symptom score = greater degree of symptom severity.
Time Frame: Up to 33.8 months
Population: The PRO analysis set included all participants with baseline and at least 1 post-baseline PRO measurement in the full analysis set. Overall number analyzed is the number of participants with data available for analysis of this outcome measure at end of treatment visit.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Brigatinib | Alectinib
Number analyzed (Participants) | 37 | 40
score on a scale
  End of Treatment: Dyspnoea | 22.22 [0.0 to 88.9] | 11.11 [0.0 to 88.9]
  End of Treatment: Coughing | 33.33 [0.0 to 100.0] | 33.33 [0.0 to 66.7]
  End of Treatment: Haemoptysis | 0.00 [0.0 to 33.3] | 0.00 [0.0 to 66.7]
  End of Treatment: Sore mouth | 0.00 [0.0 to 100.0] | 0.00 [0.0 to 66.7]
  End of Treatment: Dysphagia | 0.00 [0.0 to 100.0] | 0.00 [0.0 to 66.7]
  End of Treatment: Peripheral neuropathy | 0.00 [0.0 to 66.7] | 0.00 [0.0 to 100.0]
  End of Treatment: Alopecia | 0.00 [0.0 to 33.3] | 0.00 [0.0 to 100.0]
  End of Treatment: Pain in chest | 0.00 [0.0 to 66.7] | 0.00 [0.0 to 100.0]
  End of Treatment: Pain in arm or shoulder | 0.00 [0.0 to 66.7] | 0.00 [0.0 to 100.0]
  End of Treatment: Pain in other parts | 0.00 [0.0 to 66.7] | 0.00 [0.0 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years 4 months
Description: All-cause Mortality: FAS. Serious and Other Adverse Events: Safety Analysis Set included all participants who received at least 1 dose of study drug. As per planned analysis, data for adverse events was collected per treatment groups (brigatinib and alectinib) irrespective of the dosing regimen and is presented accordingly.
Groups:
- Alectinib: Participants were administered alectinib 600 mg, capsules, orally, BID until objective disease progression per RECIST version 1.1, as assessed by the investigator, or intolerable toxicity, or up to 59.83 months.
Arm/Group | Brigatinib | Alectinib
All-Cause Mortality (participants affected / at risk) | 37/125 | 25/123
Serious Adverse Events (participants affected / at risk) | 38/125 | 24/122
Other Adverse Events (participants affected / at risk) | 122/125 | 118/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Brigatinib (N=125) | Alectinib (N=122)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/67 | 1/68 — Number of participants at risk in each arm is based on the female population in this study.
Bronchoscopy (Investigations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/67 | 0/68 — Number of participants at risk in each arm is based on the female population in this study.
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/67 | 0/68 — Number of participants at risk in each arm is based on the female population in this study.
Chest discomfort (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/67 | 1/68 — Number of participants at risk in each arm is based on the female population in this study.
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/67 | 1/68 — Number of participants at risk in each arm is based on the female population in this study.
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Nodule (General disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pelvic mass (General disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 3
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Swelling face (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib (N=125) | Alectinib (N=122)
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Alanine aminotransferase increased (Investigations) | 59 | 47
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 8 | 0
Amylase increased (Investigations) | 26 | 14
Anaemia (Blood and lymphatic system disorders) | 27 | 45
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 19
Aspartate aminotransferase increased (Investigations) | 71 | 51
Asthenia (General disorders) | 15 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 16
Bilirubin conjugated increased (Investigations) | 2 | 10
Blood alkaline phosphatase increased (Investigations) | 16 | 25
Blood bilirubin increased (Investigations) | 7 | 39
Blood bilirubin unconjugated increased (Investigations) | 2 | 7
Blood cholesterol increased (Investigations) | 8 | 3
Blood creatine phosphokinase MB increased (Investigations) | 7 | 3
Blood creatine phosphokinase increased (Investigations) | 92 | 39
Blood creatinine increased (Investigations) | 16 | 21
Blood glucose increased (Investigations) | 9 | 3
Blood insulin increased (Investigations) | 14 | 9
Blood lactate dehydrogenase increased (Investigations) | 25 | 13
Blood urea increased (Investigations) | 1 | 9
COVID-19 (Infections and infestations) | 13 | 13
Constipation (Gastrointestinal disorders) | 14 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 26
Decreased appetite (Metabolism and nutrition disorders) | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 16 | 21
Dizziness (Nervous system disorders) | 10 | 8
Dyspepsia (Gastrointestinal disorders) | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Fatigue (General disorders) | 11 | 19
Gamma-glutamyltransferase increased (Investigations) | 8 | 2
Headache (Nervous system disorders) | 23 | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 11
Hypertension (Vascular disorders) | 38 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 8
Influenza like illness (General disorders) | 9 | 9
Insomnia (Psychiatric disorders) | 7 | 6
Lipase increased (Investigations) | 29 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 20
Nasopharyngitis (Infections and infestations) | 3 | 7
Nausea (Gastrointestinal disorders) | 18 | 11
Neutrophil count decreased (Investigations) | 3 | 7
Oedema peripheral (General disorders) | 4 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 8 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 11
Pyrexia (General disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 19 | 12
Upper respiratory tract infection (Infections and infestations) | 4 | 8
Vomiting (Gastrointestinal disorders) | 13 | 12
Weight decreased (Investigations) | 11 | 3
Weight increased (Investigations) | 6 | 12
White blood cell count decreased (Investigations) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03596866/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03596866/SAP_001.pdf